CLINICAL TRIAL: NCT04161495
Title: A Phase 3 Open-Label, Multicenter Study of the Safety, Efficacy, and Pharmacokinetics of Intravenous Recombinant Coagulation Factor VIII Fc-von Willebrand Factor-XTEN Fusion Protein (rFVIIIFc-VWF-XTEN; BIVV001) in Previously Treated Patients ≥12 Years of Age With Severe Hemophilia A
Brief Title: A Phase 3 Open-label Interventional Study of Intravenous Recombinant Coagulation Factor VIII Fc-von Willebrand Factor-XTEN Fusion Protein, Efanesoctocog Alfa (BIVV001), in Patients With Severe Hemophilia A
Acronym: XTEND-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC16293; 2019-002023-15 (EudraCT Number); U1111-1223-4867 (Registry Identifier: ICTRP)
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A | interventions — BIVV001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Prophylaxis (Experimental): Participants who were on a prophylaxis treatment with a FVIII product prior to study EFC16293 including participants who rolled over from study OBS16221, received BIVV001 50 international units per kilogram (IU/kg) intravenous (IV) injection once-weekly (QW) for 52 weeks in the current study. Study OBS16221 participants with 6 months historical data on prophylaxis treatment with a marketed FVIII product prior to enrollment were analyzed as a subgroup (named as: Arm A: Historical Prophylaxis [OBS16221]) in the outcome measure analysis.
  Interventions: Biological: efanesoctocog alfa (BIVV001)
- Arm B: On-Demand Then Prophylaxis (Experimental): Participants who were on an on-demand treatment regimen with a FVIII product prior to study EFC16293, including participants who rolled over from study OBS16221, received BIVV001 50 IU/kg IV injection as an on-demand treatment (as needed for the treatment of bleeding episodes) from Week 1 to Week 26 in current study. At Week 26, participants in Arm B were switched to prophylaxis treatment, and received BIVV001 50 IU/kg, IV injection QW until Week 52.
  Interventions: Biological: efanesoctocog alfa (BIVV001)

INTERVENTIONS:
Biological: efanesoctocog alfa (BIVV001) — Pharmaceutical form: solution for injection Route of administration: IV injection

SUMMARY:
Primary Objective:

- To evaluate the efficacy of BIVV001 as a prophylaxis treatment in prophylaxis treatment arm.

Secondary Objectives:

* To evaluate the efficacy of BIVV001 as a prophylaxis treatment.
* To evaluate the efficacy of BIVV001 in the treatment of bleeding episodes.
* To evaluate BIVV001 consumption for the prevention and treatment of bleeding episodes.
* To evaluate the effect of BIVV001 prophylaxis on joint health outcomes.
* To evaluate the effect of BIVV001 prophylaxis on Quality of Life outcomes.
* To evaluate the efficacy of BIVV001 for perioperative management.
* To evaluate the safety and tolerability of BIVV001 treatment.
* To assess the pharmacokinetics (PK) of BIVV001 based on the 1-stage activated partial thromboplastin time (aPTT) and 2-stage chromogenic coagulation factor VIII (FVIII) activity assays.

DETAILED DESCRIPTION:
Participants in prophylaxis arm received a weekly prophylactic dose of BIVV001 for 52 weeks. Participants in on-demand arm received BIVV001 on demand for 26 weeks followed by a switch to weekly prophylaxis for another 26 weeks.

The Sponsor planned to perform a long-term safety trial. Enrollment in this open-label extension study would be offered to participants completing the treatment period based on eligibility criteria.

ELIGIBILITY:
Inclusion criteria:

* Participant, male or female, must be equal to or greater than 12 years of age inclusive, at the time of signing the informed consent.
* Severe hemophilia A, defined as less than (<) 1 international units per deciliter (IU/dL) (<1 percent [%]) endogenous FVIII activity as documented either by central laboratory testing at Screening or in historical medical records from a clinical laboratory demonstrating <1% FVIII coagulant activity (FVIII:C) or a documented genotype known to produce severe hemophilia A.
* Previous treatment for hemophilia A (prophylaxis or on demand) with any recombinant and/or plasma-derived FVIII, or cryoprecipitate for at least 150 exposure days.
* Current regimen included one of the following:

  * Prophylactic treatment regimen with a FVIII product or prophylactic emicizumab therapy for at least 6 months during the previous 12 months. Appropriate washout time needs to be taken into account.
  * On-demand regimen with a FVIII product with a history of at least 12 bleeding episodes in the previous 12 months or at least 6 bleeding episodes in the previous 6 months prior to study enrollment.
* On-demand participant was accepted to move to a prophylaxis treatment regimen after 26-week on-demand period.
* Willingness and ability of the participant or surrogate (a caregiver or a family member greater than or equal to [>=] 18 years of age) to complete training in the use of the study electronic Patient Diary (ePD) and to use the ePD throughout the study.
* Ability of the participant or his or her legally authorized representative (eg., parent or legal guardian) to understand the purpose and risks of the study, willing and able to comply with study requirements and provide signed and dated informed consent or assent (as applicable) and authorization to use protected health information in accordance with national and local participant privacy regulations.

Exclusion criteria:

* Clinically significant liver disease.
* Serious active bacterial or viral infection (other than chronic hepatitis or HIV) present within 30 days of screening.
* Other known coagulation disorder(s) in addition to hemophilia A.
* History of hypersensitivity or anaphylaxis associated with any FVIII product.
* Positive inhibitor results, defined as >=0.6 Bethesda unit per milliliter (BU/mL) at screening. History of a positive inhibitor test defined as >=0.6 BU/mL. Family history of inhibitors would not exclude the participant.
* Use of Emicizumab within the 20 weeks prior to screening.
* Major surgery within 8 weeks prior to screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (47):
- United States (8):
  - Investigational Site Number 920, Los Angeles, California
  - Investigational Site Number 921, Los Angeles, California
  - Investigational Site Number 911, San Diego, California
  - Investigational Site Number 917, Gainesville, Florida
  - Investigational Site Number 919, Ann Arbor, Michigan
  - Investigational Site Number 908, Lansing, Michigan
  - Investigational Site Number 906, Las Vegas, Nevada
  - Investigational Site Number 902, Seattle, Washington
- Argentina (3):
  - Investigational Site Number 136, Buenos Aires
  - Investigational Site Number 137, Buenos Aires
  - Investigational Site Number 139, Mendoza
- Australia (2):
  - Investigational Site Number 121, Perth
  - Investigational Site Number 122, Sydney
- Investigational Site Number 161, Brussels, Belgium
- Investigational Site Number 181, Campinas, Brazil
- Bulgaria (2):
  - Investigational Site Number 171, Plovdiv
  - Investigational Site Number 172, Sofia
- Canada (2):
  - Investigational Site Number 202, Hamilton
  - Investigational Site Number 205, Hamilton
- France (4):
  - Investigational Site Number 281, Brest
  - Investigational Site Number 283, Lille
  - Investigational Site Number 282, Lyon
  - Investigational Site Number 284, Marseille
- Germany (3):
  - Investigational Site Number 304, Berlin
  - Investigational Site Number 302, Bonn
  - Investigational Site Number 303, Frankfurt
- Investigational Site Number 321, Athens, Greece
- Hungary (2):
  - Investigational Site Number 312, Budapest
  - Investigational Site Number 314, Debrecen
- Italy (2):
  - Investigational Site Number 402, Milan
  - Investigational Site Number 401, Vicenza
- Japan (6):
  - Investigational Site Number 426, Kawasaki
  - Investigational Site Number 423, Kitakyushu
  - Investigational Site Number 425, Nagoya
  - Investigational Site Number 422, Nara
  - Investigational Site Number 421, Tokyo
  - Investigational Site Number 424, Tokyo
- Investigational Site Number 435, Durango, Mexico
- Investigational Site Number 641, Utrecht, Netherlands
- South Korea (3):
  - Investigational Site Number 603, Daegu
  - Investigational Site Number 600, Seoul
  - Investigational Site Number 601, Seoul
- Investigational Site Number 521, Madrid, Spain
- Taiwan (2):
  - Investigational Site Number 531, Chang-hua
  - Investigational Site Number 532, Taipei
- United Kingdom (2):
  - Investigational Site Number 581, Basingstoke
  - Investigational Site Number 581, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Susen S, Kulkarni R, Nogami K, Peyvandi F, Konkle B, Santagostino E, Khan U, Willemze A, Bystricka L, Dumont J, Chowdary P. Outcomes in participants switching from FVIII replacement therapy to efanesoctocog alfa prophylaxis in XTEND-1: a post hoc analysis. Ther Adv Hematol. 2026 Jan 20;17:20406207251398986. doi: 10.1177/20406207251398986. eCollection 2026. PMID 41583536
- [Derived] Klamroth R, von Drygalski A, Hermans C, Park YS, Chan AKC, Kupesiz A, Alvarez-Roman MT, Malec L, Santagostino E, Neill G, Bystricka L, Dumont J, Abad-Franch L, Fetita LS, Khoo L. Perioperative Management With Efanesoctocog Alfa in Patients With Haemophilia A in the Phase 3 XTEND-1 and XTEND-Kids Studies. Haemophilia. 2025 May;31(3):391-400. doi: 10.1111/hae.70017. Epub 2025 Mar 18. PMID 40099428
- [Derived] Weyand AC, Meunier S, Suzuki N, Bystricka L, Neill G, Abad-Franch L, Willemze A, Tosetto A. Treatment of Bleeding Episodes With Efanesoctocog Alfa in Previously Treated Patients With Severe Hemophilia A in the Phase 3 XTEND-1 Study. Am J Hematol. 2025 May;100(5):813-820. doi: 10.1002/ajh.27603. Epub 2025 Feb 10. PMID 39927501
- [Derived] DiBenedetti D, Neme D, Pan-Petesch B, Willemze A, Wynn T, Kragh N, Wilson A. Patient Experience With Efanesoctocog Alfa for Severe Hemophilia A: Results From the XTEND-1 Phase 3 Clinical Study Exit Interviews. Clin Ther. 2024 Dec;46(12):1016-1023. doi: 10.1016/j.clinthera.2024.09.010. Epub 2024 Oct 15. PMID 39414418
- [Derived] von Drygalski A, Chowdary P, Kulkarni R, Susen S, Konkle BA, Oldenburg J, Matino D, Klamroth R, Weyand AC, Jimenez-Yuste V, Nogami K, Poloskey S, Winding B, Willemze A, Knobe K; XTEND-1 Trial Group. Efanesoctocog Alfa Prophylaxis for Patients with Severe Hemophilia A. N Engl J Med. 2023 Jan 26;388(4):310-318. doi: 10.1056/NEJMoa2209226. PMID 36720133
- See also: EFC16293 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25242&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 51 active sites in 19 countries. A total of 170 participants were screened between 19 November 2019 to 19 March 2021, of which 11 had screen failure due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 159 participants were enrolled in this current study (EFC16293), of which 92 participants were rolled over from study OBS16221 and then subsequently enrolled and received BIVV001 in current study.
Period: Overall Study
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand Then Prophylaxis
Started | 133 | 26
Historical Prophylaxis in OBS16221 | 82 (Number of participants rolled over from study OBS16221 who were on prophylactic treatment with a marketed FVIII product for at least 6 months during OBS16221.) | 10 (Number of participants rolled over from study OBS16221 and were on treatment with a marketed FVIII product for at least 6 months during OBS16221.)
Arm B: On-demand | 0 | 26
Arm B: Prophylaxis | 0 | 26
Completed | 124 | 25
Not Completed | 9 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Prohibited concomitant medication | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Other - Unspecified | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Prophylaxis: Participants who were on a prophylaxis treatment with a FVIII product prior to study EFC16293 including participants who rolled over from study OBS16221, received BIVV001 50 IU/kg IV injection QW for 52 weeks in the current study. Study OBS16221 participants with 6 months historical data on prophylaxis treatment with a marketed FVIII product prior to enrollment were analyzed as a subgroup (named as: Arm A: Historical Prophylaxis (OBS16221) in the outcome measure analysis.
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand Then Prophylaxis | Total Title
Number analyzed (Participants) | 133 | 26 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (15.3) | 42.8 (11.7) | 35.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 132 | 26 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 29 | 0 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 71 | 26 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Estimated Annualized Bleeding Rate (ABR) in Arm A: Prophylaxis
Description: ABR is annualized number of treated bleeding episodes (BE) per participant per year. Treated Bleeding episode: any occurrence of hemorrhage that required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered less than or equal to (<=) 72 hours apart from previous injection were considered same bleeding episode. ABR=number of treated BE during efficacy period (EP)/number of days during EP*365.25. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to the study arms and treatment regimens. This outcome measure (OM) presents estimated results (i.e., results estimated by fitting negative binomial [NB] regression model on data collected during EP).
Time Frame: Baseline to Week 52
Population: Analysis was performed on full analysis set (FAS) which included all participants who received at least 1 dose of study drug. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 133
episodes per participant per year | 0.71 [0.52 to 0.97]

2. Primary Outcome: Observed Annualized Bleeding Rate in Arm A: Prophylaxis
Description: ABR is annualized number of treated bleeding episodes per participant per year. Treated Bleeding episode: any occurrence of hemorrhage that required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. ABR=number of treated bleeding episodes during EP/number of days during EP*365.25. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to the study arms and treatment regimens. This OM presents observed results (i.e., descriptive statistics values based on the data which was collected during EP).
Time Frame: Baseline to Week 52
Population: Analysis was performed on FAS population. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 133
episodes per participant per year | 0.71 (1.43)

3. Secondary Outcome: Estimated Annualized Bleeding Rate During the Efficacy Period in Arm A: Prophylaxis - Non-inferiority Analysis
Description: ABR is annualized number of treated bleeding episodes per participant per year. Treated Bleeding episode: any occurrence of hemorrhage that required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. ABR=number of treated bleeding episodes during EP/number of days during EP*365.25. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to the study arms and treatment regimens. This OM presents estimated results (i.e., results received estimated by fitting NB regression model on data collected during EP).
Time Frame: Historical prophylaxis: From 6 months (prior to entry into study EFC16293) until the day before enrollment in EFC16293; BIVV001 prophylaxis: Baseline up to Week 52 of current study EFC16293
Population: Analysis was performed on per protocol set which included all participants who had received at least one dose of study drug and did not had important protocol deviations potentially impacting efficacy. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Groups:
- Arm A: Historical Prophylaxis (OBS16221): Participants who had 6 months historical data on prophylaxis treatment (with marketed FVIII products) in study OBS16221 prior to enrollment in current study.
- Arm A: BIVV001 Prophylaxis in EFC16293: Participants who received BIVV001 50 IU/kg (prophylaxis treatment regimen) for at least 6 months in current study (EFC16293) and had at least 6 months prophylaxis treatment regimen (with marketed FVIII products) in study OBS16221 prior to enrollment in the current study.
Arm/Group | Arm A: Historical Prophylaxis (OBS16221) | Arm A: BIVV001 Prophylaxis in EFC16293
Number analyzed (Participants) | 77 | 77
episodes per participant per year | 2.99 [2.03 to 4.42] | 0.69 [0.43 to 1.12]
Statistical Analysis 1: Comparison: Arm A: Historical Prophylaxis (OBS16221) vs Arm A: BIVV001 Prophylaxis in EFC16293; Hierarchical testing framework: used to control type I error for secondary OM analyses. Statistical testing of Arm A intra-participant comparison non-inferiority continued only when estimation of previous OM was statistically significant at 0.05 level. For Arm A intra-participant comparison, mean difference and 95% confidence interval (CI) were estimated by NB regression model in which treatment (BIVV001 prophylaxis vs historical prophylaxis vs historical prophylaxis) was treated as covariate; Test type: Non-Inferiority — Non-inferiority would be established if the upper bound of the one-sided 97.5% CI was less than 4; Mean difference = -2.30, 95% CI 2-sided [-3.49 to -1.11]

4. Secondary Outcome: Observed Annualized Bleeding Rate During the Efficacy Period in Prophylaxis - Non-inferiority Analysis
Description: as for outcome 2
Time Frame: as for outcome 3
Population: Analysis was performed on per protocol set. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Arm A: Historical Prophylaxis (OBS16221) | Arm A: BIVV001 Prophylaxis in EFC16293
Number analyzed (Participants) | 77 | 77
episodes per participant per year | 2.98 (5.21) | 0.69 (1.51)

5. Secondary Outcome: Estimated Annualized Bleeding Rate During the Efficacy Period in Arm A: Prophylaxis - Superiority Analysis
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Analysis was performed on FAS population. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Arm A: Historical Prophylaxis (OBS16221) | Arm A: BIVV001 Prophylaxis in EFC16293
Number analyzed (Participants) | 78 | 78
episodes per participant per year | 2.96 [2.00 to 4.37] | 0.69 [0.43 to 1.11]
Statistical Analysis 1: Comparison: Arm A: Historical Prophylaxis (OBS16221) vs Arm A: BIVV001 Prophylaxis in EFC16293; Tested according to hierarchical testing procedure (only performed if the previous OM was statistically significant for the considered dosing regimen). For test about Arm A intra-participant comparison superiority, rate ratio and 95% CI were estimated using NB regression model in which treatment (BIVV001 prophylaxis vs historical prophylaxis) was treated as covariate; Test type: Superiority — Superiority was declared if the upper bound of the one-sided 97.5% confidence interval was less than 1; p < 0.0001, Negative binomial regression mode; Rate ratio = 0.23, 95% CI 2-sided [0.13 to 0.42]

6. Secondary Outcome: Observed Annualized Bleeding Rate During the Efficacy Period in Arm A: Prophylaxis - Superiority Analysis
Description: as for outcome 2
Time Frame: as for outcome 3
Population: Analysis was performed on FAS population. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Arm A: Historical Prophylaxis (OBS16221) | Arm A: BIVV001 Prophylaxis in EFC16293
Number analyzed (Participants) | 78 | 78
episodes per participant per year | 2.95 (5.19) | 0.68 (1.50)

7. Secondary Outcome: Change From Baseline in Hemophilia-specific Health-related Quality of Life Questionnaire for Adults (Haem-A-QOL) Physical Health Domain Score at Week 52 in Arm A: Prophylaxis
Description: Haem-A-QoL is a participant-reported questionnaire designed for adult participants (greater than or equal to [>=] 17 years of age) with hemophilia; and consisted of 46 items comprising 10 domains (physical health [5 items], feelings [4 items], view of self [5 items], sports and leisure [5 items], work and school [4 items], dealing with hemophilia [3 items], treatment [8 items], future [5 items], family planning [4 items], partnership and sexuality [3 items]). Items were rated along five response options: never, rarely, sometimes, often, or all the time. Raw score for physical health domain were transformed to a scale ranged from 0 to 100, where lower scores denoted better physical health. Change from baseline in physical Health domain score was reported in this OM.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 98
score on a scale | -6.79 (18.59)
Statistical Analysis 1: Comparison: Arm A: Prophylaxis; Testing according to hierarchical testing procedure. Only performed if previous OM [Annualized Bleeding Rate During the Efficacy Period in Prophylaxis Arm - Superiority Analysis] was statistically significant for considered dosing regimen). Least square (LS) mean difference, standard error and 95% confidence interval were estimated by mixed-effect model with repeated measures (MMRM) using visit as fixed effect and Baseline Haem-A-QOL physical health score as covariate; Test type: Superiority; p = 0.0001, Unstructured covariance matrix; An unstructured covariance matrix within a participant was used; LS mean difference = -6.74, 95% CI 2-sided [-10.13 to -3.36], Standard Error of Mean 1.71

8. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurements Information Systems (PROMIS) Pain Intensity 3a Score at Week 52 in Arm A: Prophylaxis
Description: PROMIS is a system of reliable and precise measures of participant-reported heath status. PROMIS measures cover physical, mental and social health and can be used for many chronic conditions. PROMIS - Pain Intensity - Short Form 3a consisted of 3 questions, participants reported for the intensity of pain experienced in the past 7 days. Each question had 5 responses scored between 1 (had no pain) to 5 (very severe pain). Total PROMIS pain intensity 3a score range was from 3 (no pain) to 15 (very severe pain), where higher score indicated more intense pain. Total raw score was converted into a T-score which rescaled raw score into standardized score with mean of 50 and standard deviation (SD) of 10. Higher PROMIS T-score represented worst outcome. For PROMIS pain intensity 3a, T-score of 60 was one SD worse than average.
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 119
T-score | -1.97 (7.86)
Statistical Analysis 1: Comparison: Arm A: Prophylaxis; Testing according to hierarchical testing procedure. Only performed if previous OM [Change From Baseline in Haem-A-QOL Physical Health Score at Weeks 26 and 52: Prophylaxis Arm] was statistically significant for considered dosing regimen). LS mean difference, standard error and 95% confidence interval were estimated by MMRM using visit as fixed effect and PROMIS Pain Intensity 3a score as covariate; Test type: Superiority; p = 0.0042, Unstructured covariance matrix; An unstructured covariance matrix within a participant was used; LS mean difference = -1.94, 95% CI 2-sided [-3.26 to -0.63], Standard Error of Mean 0.67

9. Secondary Outcome: Change From Baseline in Hemophilia Joint Health Score (HJHS) Total Score at Week 52 in Arm A: Prophylaxis
Description: HJHS is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. It comprised an evaluation of the elbows, knee and ankle joints: swelling (0 to 3), duration of swelling (0 and 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2) and strength (0 to 4), in each item 0 = none and higher score = severe damage and global gait (walking, stairs, running, hopping on 1 leg) scored on scale ranged from 0 to 4, where 0 = all skills in normal limit and 4 = no skills within normal limits). Total HJHS score = sum of joint totals (0 to 120) + general gait (1 to 4) and ranged from 0 (no joint damage) to 124 (severe joint damage), where higher score indicated severe joint damage.
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 107
score on a scale | -1.5 (6.4)
Statistical Analysis 1: Comparison: Arm A: Prophylaxis; Testing according to hierarchical testing procedure (only performed if previous OM [Change From Baseline in PROMIS Pain Intensity 3a First Item at Week 52: Prophylaxis Arm] was statistically significant for considered dosing regimen). LS mean difference, standard error and 95% confidence interval were estimated by MMRM using visit as fixed effect and Baseline Haem-A-QOL physical health score as covariate; Test type: Superiority; p = 0.0101, Unstructured covariance matrix — An unstructured covariance matrix within a participant was used; LS mean difference = -1.54, 95% CI 2-sided [-2.70 to -0.37], Standard Error of Mean 0.59

10. Secondary Outcome: Annualized Bleeding Rate by Type of Bleed (Spontaneous, Traumatic and Unknown Type)
Description: ABR: annualized number of treated bleeding episodes per participant per year. EP reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. Treated bleeding episode: episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection. Spontaneous bleeding: bleeding episode without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic bleeding: bleeding episode with known/believed reason for bleed.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: Analysis was performed on FAS. Data for this OM was planned to be collected and analyzed separately in Arm B for participants during on-demand treatment and during prophylaxis treatment post switch.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Groups:
- Arm B: On-Demand: Participants who were on an on-demand treatment regimen with a FVIII product prior to study EFC16293 including participants who rolled over from study OBS16221, received BIVV001 50 IU/kg IV injection as an on-demand treatment (as needed for the treatment of bleeding episodes) from Week 1 to Week 26 in current study.
- Arm B: Prophylaxis: Participants who received BIVV001 50 IU/kg IV injection as an on-demand treatment from Week 1 to Week 26 and were switched to prophylaxis dosing and received BIVV001 50 IU/kg, IV injection QW until Week 52 in the current study.
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
episodes per participant per year
  Spontaneous | 0.00 [0.00 to 0.00] | 16.69 [8.64 to 23.76] | 0.00 [0.00 to 0.00]
  Traumatic | 0.00 [0.00 to 0.00] | 3.95 [0.00 to 6.48] | 0.00 [0.00 to 0.00]
  Unknown type | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

11. Secondary Outcome: Annualized Bleeding Rate by Location of Bleed (Joint, Muscle, Internal and Skin/Mucosa)
Description: ABR: annualized number of treated bleeding episodes per participant per year. Efficacy period reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. Treated bleeding episode: episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection. Spontaneous bleeding: bleeding episode without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic bleeding: bleeding episode with known/believed reason for bleed.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
episodes per participant per year
  Joint | 0.00 [0.00 to 1.02] | 18.42 [10.80 to 23.90] | 0.00 [0.00 to 0.00]
  Muscle | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 0.00]
  Internal | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Skin/mucosa | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 0.00]

12. Secondary Outcome: Annualized Bleeding Rate for All Bleeding Episodes
Description: ABR: annualized number of all bleeding (treated and untreated) episodes/participant/year. ABR = number of all bleeding episodes during EP/number of days in EP*365.25. EP reflects sum of all time intervals during which participants were treated with BIVV001 according to study arms and treatment regimens. Bleeding episode: episode started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any bleed at different location: considered as separate bleeding episode, regardless of time from last injection. Spontaneous: bleeding without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic: bleeding with known/believed reason.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: Analysis was performed on FAS population. Data for this OM was planned to be collected and analyzed separately in Arm B for participants during on-demand treatment and during prophylaxis treatment post switch.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
episodes per participant per year | 0.00 [0.00 to 1.15] | 21.13 [16.80 to 27.13] | 0.00 [0.00 to 1.93]

13. Secondary Outcome: Annualized Bleeding Rate: Intra-participant Comparison of Arm B Participants
Description: ABR is annualized number of treated bleeding episodes per participant per year. Treated Bleeding episode: any occurrence of hemorrhage that required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. ABR = (Number of treated bleeding episodes during EP/number of days during EP*365.25. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to the study arms and treatment regimens.
Time Frame: Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: Analysis was performed on FAS population. In this OM, ABR of Arm B: separately for participants during prophylaxis treatment versus On-Demand treatment was reported.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 26 | 26
episodes per participant per year | 21.13 [15.12 to 27.13] | 0.00 [0.00 to 0.00]

14. Secondary Outcome: Percentage of Participants Achieving Factor VIII (FVIII) Activity Levels Above 1%, 5%, 10%, 15%, and 20% in Arm A: Prophylaxis
Description: FVIII activity level was measured using activated partial thromboplastin time (aPTT)-based one stage clotting assay. Percentage of participants who achieved steady-state trough FVIII activity levels above (>) 1%, 5%, 10%, 15%, and 20% were reported for Arm A: Prophylaxis in this OM. Participants were counted in more than one row, as applicable.
Time Frame: Baseline to Week 52
Population: Analysis was performed on pharmacokinetic (PK) analysis set which included participants who had completed adequate blood sample collection to assess key PK parameters. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 131
percentage of participants
  >1% | 100
  >5% | 99.0
  >10% | 83.5
  >15% | 40.8
  >20% | 17.5

15. Secondary Outcome: Number of Injections of BIVV001 Required to Treat a Bleeding Episode
Description: The number of injections required to resolve each bleeding episode was averaged across all bleeding episodes per participant. A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was planned to be collected and analyzed separately in Arm B for participants during on-demand treatment and during prophylaxis treatment post switch.
Measure: Median (Inter-Quartile Range); unit: injections per participant
Groups:
- Arm A: Prophylaxis: Participants who were on a prophylaxis treatment with a FVIII product prior to study EFC16293 including participants who rolled over from study OBS16221, received BIVV001 50 IU/kg IV injection QW for 52 weeks in the current study. Study OBS16221 participants with 6 months historical data on prophylaxis treatment with a marketed FVIII product prior to enrollment were analyzed as a subgroup (named as: Arm A: Historical Prophylaxis [OBS16221]) in the outcome measure analysis.
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 47 | 26 | 6
injections per participant | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

16. Secondary Outcome: Total Dose of BIVV001 Required to Treat Bleeding Episode
Description: The total dose (IU/kg) used to resolve each bleeding episode was averaged across all bleeding episodes per participant. A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this OM and 'overall number of units analyzed' = total number of treated bleeding episodes. Data for this OM was planned to be collected and analyzed separately in Arm B for participants during on-demand treatment and during prophylaxis treatment post switch.
Measure: Median (Inter-Quartile Range); unit: IU/kg
Units Other Than Participants: Treated bleeding episode
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 47 | 26 | 6
Number analyzed (Treated bleeding episode) | 86 | 268 | 8
IU/kg | 50.85 [41.69 to 52.08] | 50.96 [50.10 to 51.83] | 49.79 [40.54 to 50.60]

17. Secondary Outcome: Percentage of Bleeding Episodes Treated With a Single Injection of BIVV001
Description: A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode. Percentage of bleeding episodes (of all bleeding episodes occurred) which were treated with single injection was reported in this OM.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 16
Measure: Number; unit: percentage of bleeding episodes
Units Other Than Participants: Treated bleeding episode
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 47 | 26 | 6
Number analyzed (Treated bleeding episode) | 86 | 268 | 8
percentage of bleeding episodes | 94.2 | 97.4 | 100

18. Secondary Outcome: Percentage of Participants With Response to BIVV001 Treatment Based on the International Society on Thrombosis and Haemostasis (ISTH) 4-point Response Scale
Description: The participant's response related to each injection of BIVV001 treatment for treating a bleed was evaluated using ISTH 4-point response scale categorized as: Excellent (complete pain relief/complete resolution of signs of bleeding), Good (significant pain relief/improvement in signs of bleeding), Moderate (modest pain relief/improvement in signs of bleeding) and none (no or minimal improvement/condition worsened). Assessment was performed approximately 72 hours after the initial treatment for the bleeding episode. Bleeding episode was defined as an episode that started from first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location or injections <=72 hours apart were considered same bleeding episode. Participants were counted in more than one row, as applicable.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 47 | 26 | 6
percentage of participants
  Excellent or Good | 82.2 | 98.4 | 100
  Excellent | 53.4 | 76.5 | 83.3
  Good | 28.8 | 22.0 | 16.7
  Moderate | 13.7 | 1.6 | 0
  None | 4.1 | 0 | 0

19. Secondary Outcome: Physicians' Global Assessment of Participant's Response to BIVV001 Treatment
Description: Physicians assessed participant's response to BIVV001 treatment using 4-point response scale: Excellent=bleeding episodes (BE) responded to fewer than/usual number of injections/less than/usual dose of FVIII/rate of breakthrough bleeding during prophylaxis was <= that usually observed; Effective = most BE responded to same number of injections and dose, but some required more injections/higher doses/there was minor increase in rate of breakthrough bleeding; partially effective = BE most often required more injections and/or higher doses than expected/adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses; Ineffective = routine failure to control hemostasis or hemostatic control required additional agents. Percentages were based on total number of responses.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 12
Measure: Number; unit: percentage of responses
Units Other Than Participants: Total responses
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
Number analyzed (Total responses) | 622 | 77 | 44
percentage of responses
  Excellent | 95.7 | 96.1 | 93.2
  Effective | 4.3 | 3.9 | 6.8
  Partially effective | 0 | 0 | 0
  Ineffective | 0 | 0 | 0

20. Secondary Outcome: Total Annualized BIVV001 Consumption Per Participant
Description: Total annualized BIVV001 consumption (in IU/kg) was calculated for each participant as: Total IU/kg of BIVV001 during EP divided by total number of days during EP*365.25. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to the study arms and treatment regimens.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 12
Measure: Median (Full Range); unit: IU/kg per participant per year
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
IU/kg per participant per year | 2756.99 [2385.1 to 50171.7] | 1212.27 [435.9 to 2023.8] | 2737.53 [2486.4 to 2924.8]

21. Secondary Outcome: Change From Baseline in Hemophilia Joint Health Score (HJHS) Domain Score at Week 52 in Arm A: Prophylaxis
Description: HJHS is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. Following domains were assessed for elbows, knee and ankle joints: swelling (score 0 = no swelling to 3=severe), duration of swelling (score 0 = no swelling and 1 = >=6 months), muscle atrophy (score 0 = none to 2 = severe), crepitus on motion (score 0 = none to 2=severe), flexion loss (score 0 = <5' to 3 = >20'), extension loss (score 0 = <5' to 3 = >20'), joint pain (score 0 = no pain through active range of motion to 2 = pain through active range) and strength (score 0 = holds test position with maximum resistance to 4 = trace/no muscle contraction), in each item 0 = none and higher score = severe damage.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 133
score on scale
  Swelling: number analyzed (Participants) | 114
  Swelling | -0.3 (1.2)
  Duration Of Swelling: number analyzed (Participants) | 113
  Duration Of Swelling | -0.2 (0.8)
  Muscle Atrophy: number analyzed (Participants) | 116
  Muscle Atrophy | -0.3 (1.2)
  Crepitus On Motion: number analyzed (Participants) | 114
  Crepitus On Motion | -0.3 (1.2)
  Flexion Loss: number analyzed (Participants) | 112
  Flexion Loss | -0.3 (1.6)
  Extension Loss: number analyzed (Participants) | 113
  Extension Loss | -0.2 (1.5)
  Joint Pain: number analyzed (Participants) | 114
  Joint Pain | -0.1 (1.2)
  Strength: number analyzed (Participants) | 113
  Strength | 0.3 (0.6)

22. Secondary Outcome: Estimated Annualized Joint Bleeding Rate (AJBR)
Description: AJBR: annualized number of joint bleeding/participant/year. ABR = number of treated joint bleeding episodes during EP divided by total number of days during EP*365.25. Joint bleeding episode: an unusual sensation in joint ('aura') in combination with 1) increasing swelling/warmth over skin, joint; 2) increasing pain or 3) progressive loss of range of motion or difficulty in using limb as compared with Baseline. Bleeding episode (BE): episode that started from first sign of bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location/injections <=72 hours apart were considered same bleeding episode. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: joint BE per participant per year
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
joint BE per participant per year | 0.51 [0.36 to 0.72] | 17.48 [14.88 to 20.54] | 0.62 [0.25 to 1.52]

23. Secondary Outcome: Observed Annualized Joint Bleeding Rate (AJBR)
Description: AJBR: annualized number of joint bleeding/participant/year. ABR = number of treated joint bleeding episodes during EP divided by total number of days during EP*365.25. Joint bleeding episode: unusual sensation in joint ('aura') with 1) in combination with increasing swelling/warmth over skin, joint; 2) increasing pain or 3) progressive loss of range of motion or difficulty in using limb as compared with Baseline. BE: episode that started from first sign of bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location/injections <= 72 hours apart were considered same bleeding episode. EP reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: joint BE per participant per year
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
joint BE per participant per year | 0.52 (1.09) | 17.45 (7.31) | 0.61 (1.33)

24. Secondary Outcome: Total Number of Target Joint Resolved in Participants at Week 52 in Arm A: Prophylaxis
Description: A target joint at baseline was defined as a major joint with >=3 spontaneous bleeding episodes in a consecutive 6 month period prior to entry to the study, captured at Baseline. A target joint resolved was defined as <=2 spontaneous bleeds into that joint during 12 months of continuous exposure. Total number of target joints resolved at Week 52 were reported.
Time Frame: Week 52
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this OM and 'overall number of units analyzed' = total number of evaluable target joints with >=3 spontaneous bleeding at Baseline and with 12 months continuous exposure. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Number; unit: Target joints resolved
Units Other Than Participants: Total number of evaluable target joints
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 14
Number analyzed (Total number of evaluable target joints) | 45
Target joints resolved | 45

25. Secondary Outcome: Change From Baseline in Hemophilia-specific Health-related Quality of Life Questionnaire for Adults Total Score at Week 52 in Arm A: Prophylaxis
Description: Haem-A-QoL: participant-reported questionnaire designed for adult participants (>=17 years of age) with hemophilia; and consisted of 46 items comprising 10 domains (physical health [5 items], feelings [4 items], view of self [5 items], sports and leisure [5 items], work and school [4 items], dealing with hemophilia [3 items], treatment [8 items], future [5 items], family planning [4 items], partnership and sexuality [3 items]). Items were rated along 5 response options: 1=never, 2=rarely, 3=sometimes,4=often, and 5=all the time and higher scores represent greater impairment. Raw score for each domain were transformed to a scale ranged between 0 and 100, where lower scores denoted better physical health. Haem-A-QoL Total Score was average of all domain scores and ranged from 0 to 100, where lower scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 98
score on scale | -4.56 (11.15)

26. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurements Information Systems Short Form (PROMIS-SF) Physical Function (PF) 6b at Week 52 in Arm A: Prophylaxis
Description: PROMIS-SF v2.0 PF 6b consisted of 2-items from item-improved Health Assessment Questionnaire (HAQ) and 4-items from item-improved Physical Function-10 (PF-10) instruments. Both of these instruments assessed participant's present abilities and had 5-response options: HAQ: 1=without any difficulty, 2=with little difficulty, 3=with some difficulty, 4=with much difficulty,5=unable to do and PF-10: 1=not at all, 2=very little, 3=somewhat, 4=quite a lot, 5=cannot do. Total score of PROMIS-SF PF 6b: average scores of component items, which ranged from 0 (no disability) to 100 (worst disability). T-score rescales raw scale score (sum of scores from all questions answered) into a standardized score with a mean of 50 and standard deviation of 10, based on scoring tables provided in PROMIS Scoring Manuals. Higher PROMIS T-score=more of concept being measured.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was not planned to be collected and analyzed for Arm B.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm A: Prophylaxis
Number analyzed (Participants) | 97
T-score | 0.62 (4.77)

27. Secondary Outcome: Investigators' or Surgeons' Assessment of Participant's Hemostatic Response to BIVV001 Treatment
Description: The Investigators/Surgeons who complete the surgical procedures assess the participant's response to surgery with BIVV001 treatment using a 4-point scale, where responses were categorized as worst response: 1 = Excellent, 2 = Good, 3 = Fair, and 4 = Poor/none. Higher score indicated worst response. This assessment was performed 24 hours after the surgery. A surgery can be counted in more than one response category.
Time Frame: Baseline to Week 52
Population: Analyzed on a surgery subgroup population which included all participants who had undergone major surgery after the 1st dose of study drug. Here, 'overall number of participants analyzed' = participants with major surgeries during the treatment regimen and 'overall number of units analyzed' = number of major surgeries during the treatment regimen occurred in participants analyzed.
Measure: Number; unit: major surgeries
Units Other Than Participants: Number of major surgeries
Groups:
- Participants With Major Surgery: Participant (who had at least 6 days of exposure to BIVV001) from any arm (Arm A or Arm B) who underwent major surgery (defined as any invasive operative procedure that required any of the following: opening into a major body cavity [e.g., abdomen, thorax, skull]; operation on a joint; removal of an organ; dental extraction of any molar teeth or greater than or equal to (>=) 3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier [e.g., pleura, peritoneum, dura]) after the first dose of study drug during the current study.
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 11
Number analyzed (Number of major surgeries) | 12
major surgeries
  Excellent or Good | 12
  Excellent | 12
  Good | 0
  Fair | 0
  Poor/none | 0

28. Secondary Outcome: Number of Injections Per Surgery Required to Maintain Hemostasis During Perioperative Period for Major Surgery
Description: Perioperative period was time lapse surrounding the surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). The number of injections to maintain hemostasis (a process to prevent and stop bleeding from a blood vessel) per surgery included all injections from loading dose (i.e., the preoperative injection, administered either on the day of surgery or one day prior to the surgery), to the end of surgery. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: During the perioperative period (any time during Baseline up to Week 52)
Population: Analysis was performed on surgery subgroup population. Here, 'overall number of participants analyzed' = participants with major surgeries during the treatment regimen and 'overall number of units analyzed' = number of major surgeries during the treatment regimen occurred in participants analyzed.
Measure: Number; unit: injections
Units Other Than Participants: Number of major surgeries
Groups:
- Participants With Major Surgery: Participants (who had at least 6 days of exposure to BIVV001) from any arm (Arm A or Arm B) who underwent major surgery (defined as any invasive operative procedure that required any of the following: opening into a major body cavity [e.g., abdomen, thorax, skull]; operation on a joint; removal of an organ; dental extraction of any molar teeth or greater than or equal to (>=) 3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier [e.g., pleura, peritoneum, dura]) after the first dose of study drug during the current study.
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 11
Number analyzed (Number of major surgeries) | 12
injections
  Zero injection | 1
  One injection | 11
  Two injection | 0
  Three injection | 0
  Four injection | 0
  >Four injection | 0

29. Secondary Outcome: Total Dose Required to Maintain Hemostasis From Day -1 to Day 0 During Perioperative Period for Major Surgery
Description: Perioperative period was time lapse surrounding surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). Total dose (IU/kg) was the sum across all injections per major surgery (including loading dose) needed to maintain hemostasis (a process to prevent and stop bleeding from a blood vessel) during surgery. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura). Day 0 was defined as the surgery day. The loading dose for a given surgery was the preoperative injection, administered either on the day of surgery or one day prior to the surgery (i.e., Day -1).
Time Frame: Day -1 to Day 0 (day of surgery)
Population: Analysis was performed on surgery subgroup population. Here, 'overall number of participants analyzed' = participants with major surgeries during the treatment regimen and 'overall number of units analyzed' = number of major surgeries for which a loading dose was given on the day of surgery or one day prior to surgery (i.e. Day -1).
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 11
Number analyzed (Number of major surgeries) | 11
IU/kg | 41.65 (15.21)

30. Secondary Outcome: Total BIVV001 Consumption From Day -1 to 14 During Perioperative Period for Major Surgery
Description: Perioperative period: time lapse surrounding surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). Total BIVV001 consumption were summarized from the loading dose (the day before surgery, i.e, on Day -1) up to 2 weeks following the surgery (i.e., Day 14) and were reported in this OM.
Time Frame: Day -1 to Day 14
Population: Analysis was performed on surgery subgroup population. Here, overall number of participants analyzed = participants with major surgeries during the treatment regimen and 'overall number of units analyzed' field = number of major surgeries with BIVV001 administration within Day -1 to Day 14.
Measure: Mean (Standard Deviation); unit: IU/kg per major surgery
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 11
Number analyzed (Number of major surgeries) | 12
IU/kg per major surgery | 166.71 (72.48)

31. Secondary Outcome: Number of Blood Component Transfusions Used During Perioperative Period for Major Surgery
Description: The perioperative period was the time lapse surrounding the surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). The number of blood component transfusions used during perioperative period were summarized categorically (0, 1, 2, 3 and >3) for all major surgeries for the surgery subgroup. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: During the perioperative period (any time during Baseline up to Week 52)
Population: Analysis was performed on surgery subgroup population. Here, overall number of participants analyzed = participants with major surgeries during the treatment regimen and 'overall number of units analyzed' = number of major surgeries during the treatment regimen occurred in participants analyzed.
Measure: Number; unit: transfusions per surgery
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 11
Number analyzed (Number of major surgeries) | 12
transfusions per surgery
  Zero | 12
  One | 0
  Two | 0
  Three | 0
  >Three | 0

32. Secondary Outcome: Type of Blood Component Transfusions Used During Perioperative Period for Major Surgery
Description: The perioperative period was the time lapse surrounding the surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). The type of blood component (Red blood cell, platelet, fresh frozen plasma, whole blood and other) transfusions used were summarized for all major surgeries. Post-operative referred to the day following the end of surgery to the date of hospital discharge. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: During the perioperative period (any time during Baseline up to Week 52)
Population: as for outcome 31
Measure: Number; unit: transfusions per surgery
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 11
Number analyzed (Number of major surgeries) | 12
transfusions per surgery
  Red Blood Cell | 0
  Platelet | 0
  Fresh Frozen Plasma | 0
  Whole Blood | 0
  Other | 0

33. Secondary Outcome: Estimated Blood Loss During Major Surgery
Description: The estimated total blood loss (in milliliters) during major surgeries were summarized. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: Day 0 (i.e., day of surgery)
Population: Analysis was performed on surgery subgroup population. Here, overall number of participants analyzed = participants with reported blood loss during major surgery and 'overall number of units analyzed' = number of major surgeries with blood loss report during the treatment regimen occurred in participants analyzed.
Measure: Mean (Standard Deviation); unit: milliliters
Units Other Than Participants: number of major surgery with blood loss
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 5
Number analyzed (number of major surgery with blood loss) | 6
milliliters | 143.33 (189.38)

34. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug which did not necessarily have a causal relationship with the treatment. A serious AE (SAE) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was a medically important event. Treatment-emergent AEs were AEs that developed, worsened or became serious from Baseline (Day 1) up to 3 weeks post last dose.
Time Frame: Arm A: From Baseline (Day 1) up to 3 weeks post last dose of BIVV001 (i.e., up to Week 55); Arm B: On-demand: Baseline to Week 26 and Arm B: Prophylaxis: From Week 26 up to 3 weeks post last dose of BIVV001 in Week 52 (i.e., up to Week 55)
Population: Analysis was performed on safety population which included all participants who received at least one dose of study drug. Data for this OM was planned to be collected and analyzed separately in Arm B for participants during on-demand treatment and during prophylaxis treatment post switch.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
Participants
  TEAE | 108 | 12 | 8
  TESAE | 13 | 2 | 0

35. Secondary Outcome: Number of Participants With Neutralizing Antibodies (Development of Inhibitors) Directed Against Factor VIII
Description: Development of inhibitors was defined as an inhibitor result of >=0.6 bethesda unit per milliliter (BU/mL) that was confirmed by a second test result of >=0.6 BU/mL from a separate sample, drawn 2 to 4 weeks following the date when the original sample was drawn. Both tests must have been performed by the central laboratory using the Nijmegen-modified Bethesda assay.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: Analysis was performed on safety population. Data for this OM was planned to be collected and analyzed separately in Arm B for participants during on-demand treatment and during prophylaxis treatment post switch.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
Participants | 0 | 0 | 0

36. Secondary Outcome: Number of Participants With Occurrence of Embolic and Thrombotic Events
Description: Embolic and thrombotic events were defined as arterial or venous thrombosis, confirmed by imaging.
Time Frame: Arm A: Baseline to Week 52; Arm B: On-demand - Baseline to Week 26, Prophylaxis - Week 26 to 52
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand | Arm B: Prophylaxis
Number analyzed (Participants) | 133 | 26 | 26
Participants | 0 | 0 | 0

37. Secondary Outcome: Pharmacokinetics (PK): Maximum FVIII Activity (Cmax)
Description: Cmax was defined as the maximum observed plasma FVIII Activity.
Time Frame: Baseline (15 minutes post-dose on Day 1) and 15 minutes post-dose on Week 52
Population: Analysis was performed on PK population which included all participants who had completed adequate blood sample collection to assess key PK parameters. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: IU per deciliter
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand Then Prophylaxis
Number analyzed (Participants) | 133 | 26
IU per deciliter
  Baseline | 125.05 (31.72) | 138.36 (48.66)
  Week 52: number analyzed (Participants) | 125 | 23
  Week 52 | 144.72 (36.65) | 149.42 (29.63)

38. Secondary Outcome: Pharmacokinetics: Elimination Half-life (t1/2z)
Description: Plasma t1/2z was the time measured for the plasma concentration of drug to decrease by one half. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Baseline and at Week 26; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: pre-dose, 0.25, 3, 24, 72, 168, 240 and 336 hours post-dose on Day 1 (Baseline); pre-dose, 0.25, 3, 24, 72, 168, 240, and 336 hours post-dose on Week 26
Population: Analysis was performed on PK population. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was planned to be collected and analyzed for combined population of Arm A and B. For Week 26, PK samples were collected and analyzed for arm A only as per protocol.
Measure: Median (Full Range); unit: hours
Groups:
- BIVV001 (Efanesoctocog Alfa): All participants who were enrolled in study and received BIVV001 in either Arm A or B.
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 159
hours
  Baseline | 46.5 [29.1 to 104]
  Week 26: number analyzed (Participants) | 17
  Week 26 | 46.7 [29.4 to 63.5]

39. Secondary Outcome: Pharmacokinetics: Clearance (CL)
Description: CL is defined as the rate at which the drug is removed from the body. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Baseline; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: Pre-dose, 0.25, 3, 24, 72, 168, 240 and 336 hours post-dose on Day 1 (Baseline)
Population: Analysis was performed on PK population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was planned to be collected and analyzed for combined population of Arm A and B.
Measure: Mean (Standard Deviation); unit: milliliter per hour per kilogram
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 153
milliliter per hour per kilogram | 0.508 (0.124)

40. Secondary Outcome: Pharmacokinetics: Total Clearance at Steady State (CLss)
Description: CLss is defined as the rate at which the drug is removed from the body at steady state. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Week 26; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: Pre-dose, 0.25, 3, 24, 72, 168, 240, and 336 hours post-dose on Week 26
Population: Analysis was performed on PK population. Here, 'overall number of participants analyzed' = participants with available data for this OM. Data for this OM was planned to be collected and analyzed for combined population of Arm A and B. For Week 26, PK samples were collected and analyzed for arm A only as per protocol.
Measure: Mean (Standard Deviation); unit: milliliter per hour per kilogram
Groups:
- BIVV001 (Efanesoctocog Alfa): Participants who were enrolled in sequential PK subgroup of study and received BIVV001 in Arm A or B.
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 17
milliliter per hour per kilogram | 0.449 (0.101)

41. Secondary Outcome: Pharmacokinetics: Accumulation Index (AI)
Description: AI is the ratio of accumulation of a drug under steady state conditions (i.e., after repeated administration) as compared to a single dose. AI was calculated as ratio of area under the curve (AUC) at Week 26 (Day 183) divided by AUC at Day 1, where AUC is the area under the plasma concentration versus time curve from time 0 to infinity. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Week 26; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: Pre-dose, 0.25, 3, 24, 72, 168, 240, and 336 hours post-dose on Week 26
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 15
ratio | 1.17 (0.160)

42. Secondary Outcome: Pharmacokinetics: Area Under the Plasma FVIII Activity Versus Time Curve (AUC0-tau)
Description: AUC0-tau was defined as area under the plasma concentration-time profile from time zero (pre-dose) to dosing interval. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Baseline and at Week 26; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: Pre-dose, 0.25, 3, 24, 72, 168, 240 and 336 hours post-dose on Day 1 (Baseline); pre-dose, 0.25, 3, 24, 72, 168, 240, and 336 hours post-dose on Week 26 (Day 183)
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: hour*IU/deciliter
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 159
hour*IU/deciliter
  Baseline: number analyzed (Participants) | 153
  Baseline | 9600 (2010)
  Week 26: number analyzed (Participants) | 17
  Week 26 | 11800 (2720)

43. Secondary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution (Vd) is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is the apparent volume of distribution at steady-state. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Baseline and at Week 26; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: as for outcome 42
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: milliliters per kilogram
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 159
milliliters per kilogram
  Baseline: number analyzed (Participants) | 153
  Baseline | 31.7 (7.44)
  Week 26: number analyzed (Participants) | 17
  Week 26 | 29.6 (8.26)

44. Secondary Outcome: Pharmacokinetics: Mean Residence Time (MRT)
Description: MRT is the average total time a drug molecule spends in the body. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Baseline and at Week 26; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: as for outcome 42
Population: as for outcome 38
Measure: Median (Full Range); unit: hours
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 159
hours
  Baseline: number analyzed (Participants) | 153
  Baseline | 61.9 [34.3 to 111]
  Week 26: number analyzed (Participants) | 17
  Week 26 | 66.1 [46.7 to 92.3]

45. Secondary Outcome: Pharmacokinetics: Incremental Recovery (IR)
Description: IR was calculated as (Peak activity [in IU/dL] - Trough activity [in IU/dL])/Actual Dose (in IU/kg), and peak activity at each visit was the highest activity level after the dosing, and trough activity at each visit was the activity level prior to the dosing.
Time Frame: Pre-dose, 0.25 hours post-dose on Day 1 (Baseline); pre-dose, 0.25 hours post-dose on Week 26 (Day 183)
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 159
IU/dL per IU/kg
  Baseline | 2.60 (0.648)
  Week 26: number analyzed (Participants) | 17
  Week 26 | 3.05 (0.592)

46. Secondary Outcome: Pharmacokinetics: Trough Concentration for BIVV001 (Ctrough)
Description: Ctrough is the pre-dose concentration of a drug.
Time Frame: Pre-dose at Baseline (Day 1) and Week 52
Population: Analysis was performed on PK population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Arm A: Prophylaxis | Arm B: On-Demand Then Prophylaxis
Number analyzed (Participants) | 133 | 26
IU/dL
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Week 52: number analyzed (Participants) | 120 | 25
  Week 52 | 15.70 (10.72) | 21.14 (29.59)

47. Secondary Outcome: Pharmacokinetics: Time Above Predefined (10 and 40%) FVIII Activity Levels
Description: Time above predefined (10 and 40%) FVIII activity levels mean time which BIVV001 maintains above 10 IU/dL and 40 IU/dL with single dose of 50 IU/kg. Only for participants who were enrolled in sequential PK subgroup of study, PK samples were collected for all timepoints at Baseline; however, participants did not receive BIVV001 dose in week 2 and week 27.
Time Frame: Pre-dose and 0.25, 3, 24, 72, 168, 240 and 336 hours post-dose on Day 1 (Baseline)
Population: Analysis was performed on PK population. Data for this OM was planned to be collected and analyzed for combined population of Arm A and B.
Measure: Median (Full Range); unit: hours
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 159
hours
  Time to 10 IU/dL | 185 [111 to 330]
  Time to 40 IU/dL | 85.1 [44.4 to 156]

ADVERSE EVENTS:
Time Frame: Arm A: From Baseline (Day 1) up to 3 weeks post last dose of BIVV001 (i.e., up to Week 55); Arm B: On-demand: Baseline to Week 26 and Arm B: Prophylaxis: From Week 26 to 3 weeks post last dose of BIVV001 in Week 52 (i.e., up to Week 55); Overall arm: From Baseline (Day 1) up to 3 weeks post last dose of BIVV001 (i.e., up to Week 55)
Description: Reported AEs and deaths were treatment-emergent AEs that developed, worsened or became serious from Baseline (Day 1) up to 3 weeks post last dose. Analysis was performed on safety population. AE were planned to be collected and analyzed separately in Arm B for participants during on-demand and during prophylaxis and additionally analyzed and reported for all participants combined.
Groups:
- BIVV001 (Efanesoctocog Alfa): All Participants: All participants who were enrolled in study and received BIVV001 in either Arm A or B.
Arm/Group | Arm A: Prophylaxis | Arm B: On-demand | Arm B: Prophylaxis | BIVV001 (Efanesoctocog Alfa): All Participants
All-Cause Mortality (participants affected / at risk) | 0/133 | 1/26 | 0/26 | 1/159
Serious Adverse Events (participants affected / at risk) | 13/133 | 2/26 | 0/26 | 15/159
Other Adverse Events (participants affected / at risk) | 56/133 | 7/26 | 1/26 | 64/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Prophylaxis (N=133) | Arm B: On-demand (N=26) | Arm B: Prophylaxis (N=26) | BIVV001 (Efanesoctocog Alfa): All Participants (N=159)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cubital Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Ulnar Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemophilic Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cd4 Lymphocytes Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Combined Tibia-Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Central Venous Catheter Removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device Breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Prophylaxis (N=133) | Arm B: On-demand (N=26) | Arm B: Prophylaxis (N=26) | BIVV001 (Efanesoctocog Alfa): All Participants (N=159)
Headache (Nervous system disorders) | 26 (40) | 5 (5) | 1 (1) | 32 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (31) | 1 (1) | 0 (0) | 26 (32)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1) | 0 (0) | 9 (10)
Fatigue (General disorders) | 7 (8) | 0 (0) | 0 (0) | 7 (8)
Fall (Injury, poisoning and procedural complications) | 10 (11) | 0 (0) | 0 (0) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT04161495/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT04161495/SAP_001.pdf